CLINICAL TRIAL: NCT00208338
Title: A Prospective, Randomised Pilot Study to Determine the Variability of Early Clinical Outcome in Subjects Undergoing Full Thickness Rotator Cuff Tear Repair, When Augmented With or Without Porcine Small Intestine Submucosa (RESTORE)
Brief Title: Pilot Study to Evaluate the Restore Orthobiologic Implant in Rotator Cuff Tear Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT 04/17
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Arm Injuries
Keywords: Rotator cuff tear repair
MeSH Terms: conditions — Arm Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rotator cuff repair with RESTORE Porcine Small Intestine Submucosa patch (RESTORE SIS Patch) reinforcement
  Interventions: Device: RESTORE SIS Patch
- 2 (Active Comparator): Standard rotator cuff repair
  Interventions: Procedure: Rotator cuff repair

INTERVENTIONS:
Device: RESTORE SIS Patch — Surgical repair of torn rotator cuff with RESTORE Porcine Small Intestine Submucosa patch (RESTORE SIS Patch) reinforcement
  Arms: 1
Procedure: Rotator cuff repair — Standard surgical repair of torn rotator cuff
  Arms: 2

SUMMARY:
Primary Endpoints:

Comparative evaluation of any differences between the two groups in change from baseline to the 3-month time point in terms of:

* Functional recovery (patient-based) - using the Oxford Shoulder Score.
* Functional recovery and early return of strength (pain, activities of daily living [ADL], range of motion [ROM], and power) - evaluated using the Constant Shoulder Assessment.
* Functional recovery (pain and function - patient-based), evaluated using the American Shoulder and Elbow Surgeons (ASES) Shoulder Assessment - patient self-report section.
* Region-specific Quality of Life - using the Western Ontario Rotator Cuff (WORC) Index.
* Range of motion - assessed by goniometer recorded as part of the Constant Score.
* Pain (taken from Pain visual analog scale [VAS] of the ASES Shoulder Assessment); and
* Record of escape pain medication usage (recorded in a daily patient diary).

Secondary Endpoints:

Comparative evaluation of any difference between the two groups in change from baseline to the 6-week time point, in terms of:

* Pain (taken from Pain VAS of the ASES Shoulder Assessment) and record of escape pain medication usage (recorded in a daily patient diary).

Comparative evaluation of any differences between the two groups in change from baseline to the 6-month time point, in terms of:

* Functional recovery (patient-based) - using the Oxford Shoulder Score.
* Functional recovery and early return of strength (pain, ADL, ROM, and power) - evaluated using the Constant Shoulder Assessment.
* Functional recovery (pain and function - patient-based), evaluated using the ASES Shoulder Assessment - patient self-report section.
* Region-specific Quality of Life - using the Western Ontario Rotator Cuff Index.
* Range of motion - assessed by goniometer recorded as part of the Constant Score.
* Pain (taken from Pain VAS of the ASES Shoulder Assessment) and record of escape pain medication usage (recorded in a patient diary).

Comparative evaluation of any difference between the two groups in change from baseline to the 6-week, 3, 6 and 12 month time points, in terms of health status - assessed by the EQ-5D instrument.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 40 and above.
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
* Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures, and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects whose clinical symptoms and diagnosis suggest that they have a full-thickness rotator cuff tear (which includes but is not limited to the supraspinatus), which is degenerate in nature.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition that would prevent them from fulfilling the requirements of the Clinical Investigation Plan. (This should be detailed in the Screening Log.)
* Women who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical study with an investigational product in the last 6 months.
* Subjects who are currently known to be involved in any injury litigation claims relating to the shoulder being treated as part of the study.
* Subjects with a known allergy to porcine material or who, for religious or other reasons, are unwilling to accept a porcine-derived implant.
* Subjects who have undergone previous shoulder surgery (excluding purely-diagnostic arthroscopy).
* Subjects with significant paralysis of the shoulder.
* Subjects with inflammatory arthropathies.
* Subjects with active joint or systemic infection.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-07; Primary Completion 2007-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Difference demonstrated between two groups on the Oxford Shoulder Score from baseline to 3 months | 3 months
Difference demonstrated between two groups on the Constant Shoulder Assessment from baseline to 3 months | 3 months
Difference demonstrated between two groups on the ASES Shoulder Assessment from baseline to 3 months | 3 months
Difference demonstrated between two groups on the Western Ontario Rotator Cuff Index from baseline to 3 months | 3 months

SECONDARY OUTCOMES:
Difference demonstrated between the two groups on the ASES Shoulder Assessment from baseline to 6 weeks. | 6 weeks
Difference demonstrated between the two groups on the ASES Shoulder Assessment from baseline to 6 months | 6 months
Difference demonstrated between 2 groups on EQ-5D from baseline to 6 weeks | 6 weeks
Difference demonstrated between the two groups on the Constant Shoulder Assessment from baseline to 6 months | 6 months
Difference demonstrated between the two groups on the Oxford Shoulder Score from baseline to 6 months | 6 months
Difference demonstrated between the two groups on the Western Ontario Rotator Cuff from baseline to 6 months | 6 months
Difference demonstrated between 2 groups on EQ-5D from baseline to 3 months | 3 months
Difference demonstrated between 2 groups on EQ-5D from baseline to 6 months | 6 months
Difference demonstrated between 2 groups on EQ-5D from baseline to 12 months | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- U.Z. Gasthuis Berg, Leuven, Belgium
- Royal Liverpool University Hospital, Liverpool, United Kingdom